CLINICAL TRIAL: NCT04488796
Title: STAND UP to SARS-CoV-2 (COVID-19): Using Behavioural Economics to Reduce Sedentary Behaviour in At-home Office Workers, a Pilot Randomized Controlled Trial
Brief Title: STAND UP to SARS-CoV-2 (COVID-19): Using Behavioural Economics to Reduce Sedentary Behaviour in At-home Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Marc Mitchell, Dr. Marc Mitchell, Western University, Canada
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 116127
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Health Behaviour Change
Keywords: randomized controlled trial; office-workers; sedentary behaviour; mHealth; behavioural economics

STUDY DESIGN:
Intervention Model Description: This will be a 2 (automated vs. choice of automation) by 3 (Opt-in, active choice or enhanced active choice) factorial design pilot randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Assigned Strategies: Opt-in (Experimental): Participants in this group will be assigned two behavioural strategies under the theme of "moving more" and will be asked to "Place a check in the box [agree] if you will breakup your sitting throughout your work hours by X this week". The strategy statement is followed up by; OR, click the next button at the bottom." Within the opt-in condition, the default is to not participate (by clicking "next"): participants are not required to explicitly state they do not want to do the strategy
  Interventions: Behavioral: Assigned Strategies: Opt-in
- Assigned Strategies; Active Choice (Experimental): Participants in this group will be assigned two behavioural strategies under the theme of "moving more". In the Active choice condition, participants will be required to either, "Place a check in one box: I will break up my sitting throughout my work hours by [strategy] this week or, I will not break up my sitting throughout my work hours by [strategy] this week".
  Interventions: Behavioral: Assigned Strategies: Active Choice
- Assigned Strategies; Enhanced Active Choice (Experimental): Participants in this group will be assigned two behavioural strategies under the theme of "moving more". In the Enhanced Active Choice condition, participants will to required to choose between two alternatives: "I will break up my sitting throughout my work hours this week by [strategy] to reduce my risk of diabetes, mental health issues and other detrimental health outcomes and I want to win the eGiftcard or, I will not break up my sitting time during my work hours by [strategy] this week even if it means I increase my risk of developing diabetes, mental health issues and other detrimental health outcomes and I don't care about winning an eGiftcard"
  Interventions: Behavioral: Assigned Strategies: Enhanced Active Choice
- Choice of Assignment; Opt-in (Experimental): Those opting to be assigned strategies ("Choice Strategy Assignment" group) will be assigned two random strategies, just like the "No Choice Strategy Assignment" group; however, they remain different from the "No Choice Strategy Assignment" group because they were given and chose the option to be given strategies. Those selecting to choose and manage their own strategies "Choice Strategy Self-Selection" group will be presented the same ten strategies each week, in random order, and will have the option to choose two strategies. The strategies can remain the same or change from week to week.
  Interventions: Behavioral: Choice of Assignment: Opt-in
- Choice of Assignment; Active Choice (Experimental): Those opting to be assigned strategies ("Choice Strategy Assignment" group) will be assigned two random strategies, just like the "No Choice Strategy Assignment" group; however, they remain different from the "No Choice Strategy Assignment" group because they were given and chose the option to be given strategies. Those selecting to choose and manage their own strategies "Choice Strategy Self-Selection" group will be presented the same ten strategies each week, in random order, and will have the option to choose two strategies. The strategies can remain the same or change from week to week.
  Interventions: Behavioral: Choice of Assignment: Active Choice
- Choice of Assignment; Enhanced Active Choice (Experimental): Those opting to be assigned strategies ("Choice Strategy Assignment" group) will be assigned two random strategies, just like the "No Choice Strategy Assignment" group; however, they remain different from the "No Choice Strategy Assignment" group because they were given and chose the option to be given strategies. Those selecting to choose and manage their own strategies "Choice Strategy Self-Selection" group will be presented the same ten strategies each week, in random order, and will have the option to choose two strategies. The strategies can remain the same or change from week to week.
  Interventions: Behavioral: Choice of Assignment: Enhanced Active Choice

INTERVENTIONS:
Behavioral: Assigned Strategies: Opt-in — Participants will be assigned two behavioural strategies with the opt-in choice structure
  Arms: Assigned Strategies: Opt-in
Behavioral: Assigned Strategies: Active Choice — Participants will be assigned two behavioural strategies with the Active choice structure
  Arms: Assigned Strategies; Active Choice
Behavioral: Assigned Strategies: Enhanced Active Choice — Participants will be assigned two behavioural strategies with the Enhanced Active choice structure
  Arms: Assigned Strategies; Enhanced Active Choice
Behavioral: Choice of Assignment: Opt-in — Participants will have the choice to be assigned strategies or to manage their own strategies. The strategies will be assigned using the Opt-in choice structure
  Arms: Choice of Assignment; Opt-in
Behavioral: Choice of Assignment: Active Choice — Participants will have the choice to be assigned strategies or to manage their own strategies. The strategies will be assigned using the Active choice structure
  Arms: Choice of Assignment; Active Choice
Behavioral: Choice of Assignment: Enhanced Active Choice — Participants will have the choice to be assigned strategies or to manage their own strategies. The strategies will be assigned using the Enhanced Active choice structure
  Arms: Choice of Assignment; Enhanced Active Choice

SUMMARY:
In COVID-19 times, there has been a large increase in number of people working from home; with limited places to go, an abrupt change to people's lives and lack of knowledge about the dangers of sedentary behaviour (SB), it is important to help workers develop and effortlessly incorporate healthy movement routines to optimize daily productivity and health. The combined lack of knowledge on literature on SB profiles of full time, home-based workers, effects of framing of SB reduction strategies, and strategy preference uncertainty makes for a novel study. This will be a 4-week intervention that looks at whether telling a full time, home-based office worker to do pre-selected strategies using different framing structures to break up their sedentary behaviour (SB) (i.e. sitting) will change their SB profiles. Investigators are looking to see whether having the choice (or not) to choose strategies in an unfamiliar health related selection (preference uncertainty) will create greater changes in SBs. As well, the researchers are incorporating behavioural economics' by altering choice structure in relation to behaviour change and program engagement. Workers' work-related SB will be measured by a device at baseline and on the last week of the intervention. Workers will be provided with an SB educational video to increase knowledge and motivation for change. Any SB changes in relation to productivity, mental wellness, behaviour intentions etc. will also be measured.

DETAILED DESCRIPTION:
Regardless of group assignment, participants will receive the same three-minute educational video at the beginning (week 1) and halfway through (week 3) the intervention. Each group will also receive two weekly sedentary behaviour reduction strategies that align with the concept of "moving more often".

Participants will be initially randomized into the no choice strategy assignment or choice of strategy assignment groups, then immediately randomized into one of three choice structure conditions. The strategy assignment groups (no choice and choice) will receive two individually randomized (out of the ten "move more" strategies (see Table 2) each week. The two assigned strategies will be randomized to the participant each week; therefore, strategies may or may not change week to week. When presented with the two strategies, the Qualtrics program will state: "These will be your two move more strategies (click next to acknowledge you have seen your strategies)", followed by two multiple choice styled strategies. Regardless of if the person decides to click the boxes beside the strategies or clicks "next", the strategies will be inserted into the one of the three choice structure statements. Those randomized into the "choice of strategy assignment" group will be asked in their baseline questionnaire whether or not they: "prefer to choose and manage their own sitting reduction strategies from a list of expert recommended strategies OR prefer to be assigned with two strategies every week from a list of expert recommended strategies". Those opting to be assigned strategies ("Choice Strategy Assignment" group) will be assigned two random strategies, just like the "No Choice Strategy Assignment" group; however, they remain different from the "No Choice Strategy Assignment" group because they were given and chose the option to be given strategies. Those selecting to choose and manage their own strategies "Choice Strategy Self-Selection" group will be presented the same ten strategies each week, in random order, and will have the option to choose two strategies. The strategies can remain the same or change from week to week.

As mentioned, participants will be randomly assigned to one of three choice structure conditions: opt-in, Active Choice or Enhanced Active Choice. All three messages will contain the following introduction: "As you now know, breaking up your sitting every 45 minutes with 2-3 minutes of light activity can significantly reduce negative health risks associated with prolonged sitting." This message will end with one of the three choice structures.

In the opt-in condition they will be asked to "Place a check in the box [agree] if you will breakup your sitting throughout your work hours by [strategy] this week". The strategy statement is followed up by; OR, click the next button at the bottom." Within the opt-in condition, the default is to not participate (by clicking "next"); participants are not required to explicitly state they do not want to do the strategy.

In the Active choice condition, participants will be required to either, "Place a check in one box: I will break up my sitting throughout my work hours by [strategy] this week or, I will not break up my sitting throughout my work hours by [strategy] this week".

In the Enhanced Active Choice condition, participants will to required to choose between two alternatives: "I will break up my sitting throughout my work hours this week by [strategy] to reduce my risk of diabetes, mental health issues and other detrimental health outcomes and I want to win the eGiftcard or, I will not break up my sitting time during my work hours by [strategy] this week even if it means I increase my risk of developing diabetes, mental health issues and other detrimental health outcomes and I don't care about winning an eGiftcard"

Assigned or self-selected strategies (depending initial group assignment) will be sent in a reminder email on the Wednesday morning of each week and participants will be instructed to self-report their sedentary behaviour patterns on the Friday of each week.

An "interested" participant will email research personal with their initial "interest" in which the research personnel will respond by sending them the baseline questionnaire along with their unique ID code to access it in SoSci. Participants baseline questionnaires will be randomized to be either, a) assignment of choice strategies or b) choice of assignment vs self-management of choice strategies. Those assigned to the "Choice of Assigned Strategies" condition will have an additional question presenting them with the option of having strategies assigned to them or the option to choose and manage their own strategies. The LOI will be the first page of the questionnaire for them to review, and at the bottom will state, "Clicking on the "agree" button below indicates that you have read the above information, you voluntarily agree to participate and you are at least 18 years of age. If you do not wish to participate in the research study, please decline participation by clicking on the "disagree" button and simply exit the browser." Upon completion of the baseline questionnaire, participants will be emailed a PDF version of the LOI/informed consent, and will be asked to sign (digitally) the form and email it back to research personnel. Once consent is received, participants will be randomized into one of 3 choice structure conditions (Opt-in Choice OR Active Choice OR Enhanced Active Choice).

The activPAL will be sent by courier (i.e. FedEx) and participants will receive another email with detailed instructions of how to apply the device [i.e. applied to the mid-thigh using Tegaderm (3M)] along with how to contact investigators upon any issues with application. Participants will be instructed to apply the device on Sunday evening (if possible) and to wear the device all day for a period of 5 working days (Monday to Friday). Once participants complete the device measured baseline assessment, they will place the device back in the package it came in, and using pre-paid postage, the device will be picked up (via courier) and they will then be randomized into one of the three experimental conditions preceding the intervention period. Strategies will be pre-randomized for each condition from the longlist group.

Intervention Week 1. On day one of the intervention (Monday), participants will receive an email containing, 1) a link to watch a 3-minute whiteboard-styled educational video about sedentary behaviour (i.e. health consequences, benefits of breaking up or reducing sedentary behaviour, sedentary behaviour in relation to productivity and mood etc.) and 2) another link that will lead them to a short questionnaire assessing knowledge on sedentary behaviour (fidelity check) as well as their behavioural strategies (different based on the condition assignment; as described earlier). Wednesday morning, they will receive an email reminding them of their strategies. On the last day of the same workweek (Friday), participants will be prompted (via email) with a link (Soci) to self-report their sitting habits (i.e. break frequency and break duration).

Intervention Week 2. On the Monday of week 2, participants will again be assigned or asked to choose their strategies via email (depending on group allocation) for that week and will again receive an email Wednesday morning reminding them of their chosen/assigned strategies. They will again be asked to self-report their sitting habits (via link sent through email) (i.e. break frequency and break duration) on the last day of the week (Friday).

Intervention Week 3. On the Monday of Week 3, strategies will reset as earlier described for each condition. However, for this week, the participants will be reminded of the video they watched at the beginning of the intervention and be asked to re-watch the same video. In line with the same protocol described in the earlier weeks, a reminder email will be sent on Wednesday morning and self-reported sitting habits will be measured at the end of the week.

Intervention Week 4. Week four of the intervention will be the final week. Again, strategies will reset for all conditions as previously described. Participants again, will wear the activPAL4's (delivered via FedEx) for a total of five days (Monday to Friday). This will serve as the follow-up objectively (device) measured sedentary behaviour measurement. The participants will receive the same reminder email as previous weeks. This last week, however, the Friday questionnaire will include all secondary outcomes that were initially assessed at baseline along with a short exit survey asking about participant satisfaction with the intervention.

Follow Up. Follow-up will occur two weeks post-intervention. Participants will recomplete all secondary outcomes that were initially assessed at baseline (with exception to the activPAL measurements).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Self-declare working 5 days per week (Monday to Friday)
* Full-time worker/employee (i.e. employed ≥ 30 hours/week)
* Desk-based office worker currently only working from home
* Have access to a computer with Internet and email
* Able to read and write in English

Exclusion Criteria:

* Self-declared medical condition or physical limitation that prevents them from being physically active
* Planning on leaving the current employer or taking a leave of absence for more than 3 consecutive workdays for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Change in sedentary behaviour break frequency | change from baseline to 4 weeks
  measured via ActivPAL
Change in sedentary behaviour break duration | change from baseline to 4 weeks
  measured via ActivPAL

SECONDARY OUTCOMES:
Change in work-related quality of life | change from baseline to 6 weeks
  Short form 36 health survey (SF-36) measured on a 5-point Likert scale from 1 "all of the time" to 5 "None of the time".
Change in Health outcomes | change from baseline to 6 weeks
  Questions regarding work productivity, concentration and focus will be measured with questions adapted from The Health and Work Questionnaire (HWQ). The HWQ is a multidimensional tool used to measure various aspects of productivity. The HWQ consists of 24 questions, several items being multi-part questions with internal consistency scores ranging from alpha = 0.72 to 0.96. The questions are designed to assess work quality, quantity, and efficiency, as well as impatience, concentration/focus, work satisfaction and non-work satisfaction. For the current study, 15 items were chosen from this questionnaire that were relevant to "home-based" office workers. Items will be assessed with a ten-point response scale, tailored to each question (e.g., "my worst ever" to "my best ever").
Change in sitting time | change in baseline to 4 weeks
  measured with the ActivPAL4
Change in standing time | change in baseline to 4 weeks
  measured with the ActivPAL4
Change in moving time | change in baseline to 4 weeks
  measured with the ActivPAL4
Change in prolonged sitting bouts | change in baseline to 4 weeks
  measured with the ActivPAL4
Change in percentage of time spent sitting | change from baseline to 6 weeks
  The validated three-item modified Occupational Sitting and Physical activity questionnaire (OSPAQ). The OSPAQ is a brief instrument reported to have excellent test-retest reliability (intraclass correlation coefficients = 0.73-0.90), moderate criterion validity for time spent sitting and standing (r = 0.65 and 0.49, respectively), and lower validity for time spent walking (r = 0.29). At each assessment period (baseline, week 1, week 2, week 3, week 4 and follow-up), participants will be asked to record both the number of days they were at work and total number of hours they worked in the last 7 days. Participants will then be asked to record a percentage of time spent sitting, standing, and moving (i.e. walking) (cumulative total of 100%) during work hours on a typical workday in the last 7 days.
Change in percentage of time spent standing | change from baseline to 6 weeks
  The validated three-item modified Occupational Sitting and Physical activity questionnaire (OSPAQ). The OSPAQ is a brief instrument reported to have excellent test-retest reliability (intraclass correlation coefficients = 0.73-0.90), moderate criterion validity for time spent sitting and standing (r = 0.65 and 0.49, respectively), and lower validity for time spent walking (r = 0.29). At each assessment period (baseline, week 1, week 2, week 3, week 4 and follow-up), participants will be asked to record both the number of days they were at work and total number of hours they worked in the last 7 days. Participants will then be asked to record a percentage of time spent sitting, standing, and moving (i.e. walking) (cumulative total of 100%) during work hours on a typical workday in the last 7 days.
Change in percentage of time spent moving | change from baseline to 6 weeks
  The validated three-item modified Occupational Sitting and Physical activity questionnaire (OSPAQ). The OSPAQ is a brief instrument reported to have excellent test-retest reliability (intraclass correlation coefficients = 0.73-0.90), moderate criterion validity for time spent sitting and standing (r = 0.65 and 0.49, respectively), and lower validity for time spent walking (r = 0.29). At each assessment period (baseline, week 1, week 2, week 3, week 4 and follow-up), participants will be asked to record both the number of days they were at work and total number of hours they worked in the last 7 days. Participants will then be asked to record a percentage of time spent sitting, standing, and moving (i.e. walking) (cumulative total of 100%) during work hours on a typical workday in the last 7 days.
Change in sedentary break frequency | change from baseline to 6 weeks
  measured using a modified version of the SIT-Q 7d;modified the base questionnaire to include domain-specific (work-related) break frequency and duration scores, which were the only items assessed for purposes of this study
Change in sedentary break duration | change from baseline to 6 weeks
  measured using a modified version of the SIT-Q 7d;modified the base questionnaire to include domain-specific (work-related) break frequency and duration scores, which were the only items assessed for purposes of this study

CONTACTS AND LOCATIONS:
Overall Officials: Marc Mitchell, PhD, Principal Investigator — Western University
Locations (1):
- University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No